CLINICAL TRIAL: NCT03352635
Title: Mechanisms of Ethnic/Racial Differences in Lung Cancer Due to Cigarette Smoking Clinical and Biomarkers Core: Observation Study
Brief Title: Mechanisms of Ethnic/Racial Differences in Lung Cancer Due to Cigarette Smoking Clinical and Biomarkers Core
Status: Withdrawn | Type: Observational
Why Stopped: Study was completed at other sites
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 5P01CA138388-06
Record Dates: First submitted 2017-07-25; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Tobacco Use
Keywords: Ethnic Differences
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, buffy coat, and red cells; mouthwash and buccal cells samples; urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Native Hawaiians: One parent of Hawaiian descent.
- Japanese Americans: Two parents of Japanese descent.
- Non-Hispanic Whites: Two parents of non-Hispanic white descent.

SUMMARY:
The purpose of the study is to collect human biological samples and measurements from people of various ethnic and racial backgrounds for projects related to the "Mechanisms of Ethnic/Racial Differences in Lung Cancer Due to Cigarette Smoking" Program Project Grant. These samples will be used to evaluate and compare biomarkers of tobacco exposure across Japanese Americans, Whites, and Native Hawaiians and to add to the Multiethnic Cohort (MEC) biorepository to develop or assess future biomarkers.

DETAILED DESCRIPTION:
This cross-sectional, observational study will primarily recruit smokers from the MEC study. The biological samples from these smokers are being collected since they do not currently exist in the biorepository (e.g. buccal cells). Potential smokers from the three racial groups who meet specific inclusion criteria will be invited to participate in the study. Should recruitment from the MEC sample be insufficient, smokers who meet the criteria will be recruited from the general population. This study will involve one to two home visits where tobacco use and medical history and biological samples will be collected including blood, buccal cells and urine.

Approximately 300 smokers will be recruited from the Multiethnic Cohort (MEC) study or the general population in Hawai'i. 100 participants from each of the three designated ethnic/racial groups: Native Hawaiians, Japanese Americans and Non-Hispanic Whites. All participants will be recruited from Hawai'i to reduce variation due to geographical location and maximize ability to recruit the targeted ethnic/racial groups.

This study will involve one to two home visits where demographics, tobacco use and exposure history, medical history and medication use, questionnaires assessing tobacco dependence, alcohol use, and environmental exposures will be administered. and biological samples will be collected including blood, buccal cells and urine.

ELIGIBILITY:
Inclusion Criteria:

1. One of the three targeted ethnic groups: 1)Japanese American - two parents of Japanese descent; 2) Non-Hispanic Whites - two parents of non-Hispanic white descent; 3) Native Hawaiians will include individuals with at least one parent of Hawaiian descent;
2. Smoke 5 cigarettes per day over the past three months;
3. >21 years of age;
4. Consumes 14 or fewer drinks of alcohol per week;
5. Generally stable and good health (determined by review of medical history);
6. Able to provide written voluntary consent before performance of any study related procedure.

Exclusion Criteria:

1. Current use of other nicotine containing products for > 4 times per month (and no use of any nicotine-containing products except cigarettes for 2 weeks prior to their study visits);
2. Acute or uncontrolled medical or psychiatric conditions;
3. Currently taking any medications that affect relevant metabolic enzymes or anti- inflammatory medications such as ibuprofen (this will be reviewed by study investigators on a case-by-case basis);
4. Active infection (e.g., influenza, cold, respiratory infection, sinus infection) at the time of the visit;
5. Pregnant or nursing or planning on becoming pregnant during the study;
6. Unable to read and understand English.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cigarette smokers who are Japanese American, Non-Hispanic Whites - two parents of non-Hispanic white descent or Native Hawaiians over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Project 3: Analysis of 1,3-butadiene DNA adducts | Baseline
  Ethnic differences in butadiene-DNA adducts across racial groups to determine the relationship of DNA adducts to lung cancer and the influence of carcinogen metabolizing genes on DNA adduct formation, repair, and toxicity/mutagenicity.
Project 4: Correlation of DNA adducts of buccal cells and urinary markers and lung cancer risk | Baseline
  DNA adduct levels in oral cells, themselves or together with urinary biomarker levels, correlate with lung cancer risk across various ethnic/racial groups
Project 2: NNK α-hydroxylation | Baseline
  Analysis of biomarkers of NNK α-hydroxylation (bioactivation) pathway and the effect of P450 2A6 activity on this process.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PHD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Tobacco Research Programs University of Minnesota, Minneapolis, Minnesota
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Intend to share findings from this research through publications and presentations. Institutions and individuals wishing to access any resources or data must contact the Principal Investigator (Hatsukami). Data will be available in two formats. One will be a summary of the data, with graphs and tables, posted as pdf files and as raw individual-level data for analysis. Data generated by this grant will be made to outside investigators, according to NIH Guidance. When data are shared, there will be no limits placed on how the data will be used, and co-authorship is not required as a condition for receiving data. Users will agree, however, that the recipient must not transfer the data to other users and that the data are only to be used for research purposes. A record of transfer of data and a copy of the dataset that was distributed will be kept by University of Minnesota.
Supporting Information: Study Protocol
Time Frame: Data will not be available until primary papers are accepted for publication.
Access Criteria: Persons requesting data must do so in writing, identifying the affiliation and how the data will be used.